CLINICAL TRIAL: NCT05705986
Title: Immunoregulatory Effect of Microparticle Delivered STING Agonist in the Control of Experimental Autoimmune Encephalomyelitis (EAE) and Multiple Sclerosis (MS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 20D.098
Record Dates: First submitted 2021-04-20; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Relapse Remitting Multiple Sclerosis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood Draw — Single blood draw

SUMMARY:
Microparticles (MPs) as a mode of therapeutic delivery can selectively deliver immunomodulatory treatment to the phagocytic cells, particularly dendritic cells (DCs), inducing their tolerogenic phenotype and function and T regulatory (Treg) cell expansion. The study will characterize the in vitro response of cGAMP immunomodulator incapsulated microparticles on the capacity of DCs and Tregs to regulate the inflammatory response.

DETAILED DESCRIPTION:
This is a lab study only. No medication will be dispensed as a part of the study. No tests or procedures will be performed. Blood ( approximately 10 teaspoons ; 10 green top tubes) will be drawn by a qualified phlebotomist, nurse or physician in the Neurology clinic, during routine clinic visits. Proper medical procedures will be followed when collecting blood to minimize patient risk. In addition, steps will be taken to guard patient's confidentiality. Unique codes will be assigned to each sample. All identifying information will be removed from samples and clinical data before they are given to the research staff conducting the laboratory study. Only the clinic staff will have access to the consent forms, the master list (that connect the unique codes with the patient names) and subject medical records. The blood draw will coincide with the subject's regular visit to the Neurology clinic.

All records will be secured with the current PACS radiology system and computerized information systems/computerized databases which are the current methods for securing all patient information. Care will be taken to preserve the confidentiality of all patient-related information. Material with identifying information will be stored in the clinic locked data storage room. Patient names will not be used in any publications. Results of laboratory studies performed on these samples will not be shared with subjects. Laboratory results will not be incorporated into patients medical records.

The proposal states to separate dendritic cells using magnetic beads separation and use them as an antigen presenting cells to T cells.The therapeutic effect of the nanoparticle delivered phosphatidylserine (PS, PAR-PS) will be measured, using cytokine secretion and the detection of the T regulatory (Treg) cell induction. Proliferation will be determined using CFSE, cytokine secretion will be measured using ELISA and the intracellular cytokine staining for IFNg, IL-17A, IL-17F, IL-21, IL-22, TGFb, IL-10 and IL-4. The induction of Treg cells will be measured using flow cytometry and determining the percentage of CD4+ CD25+ CD127- FoxP3+ Treg cells within the CD4+ lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects meeting diagnostic criteria for relapsing remitting multiple sclerosis
2. Between the ages of 18-55
3. Not treated with immunomodulatory therapy, no other neurological diagnosis, no other inflammatory disease

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 40 patients diagnosed with relapse remitting multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Characterize cGAMP MP-induced tolerogenic DCs from RRMS patients. | Baseline
  Flow cytometry study will measure the cGAMP MP phagocytosis by PBMCs and characterize the phenotype of cGAMP MP-induced DCs of 40 untreated RRMS patients after incubation with fluorescently-labelled cGAMP MPs.
Determine the capacity of cGAMP MP-treated DCs to induce iTreg expansion in human in-vitro cultures | Baseline
  Flow cytometry studies will characterize the induced Treg phenotype generated after co-culture with cGAMP MP-treated DCs cells to determine the capacity of the cGAMP MP-treated DCs to induce differentiation and expansion of iTregs

SECONDARY OUTCOMES:
Determine the transcriptome of cGAMP MP IL-27- and IL-10-induced Tregs. | Baseline
  RNA sequencing of iTreg cells after coculture with cGAMP MP-treated (vs. blank MP-treated) DCs from 10 RRMS patients will detect the differentially expressed genes between cGAM MP- and blank MP-induced iTregs. The expression of transcription factors identified by RNAseq will be confirmed by RT-PCR and western blot, more quantitative methods.
Determine the in-vitro reconstitution of iTreg suppressive function in RRMS patients after coculture with cGAMP MP-treated DCs. | Baseline
  Suppression assay will determine to what extent Treg cells from co-cultures with cGAM-MP-treated DCs increase (restore normal) suppressive function in comparison to the co-cultures with blank MP-treated DCs.
Induction of antigen-specific immune tolerance after co-administer DR2-aAPMs with the cGAMP MPs to DCs. | Baseline
  The suppressive effect of sorted Tregs induced after co-administration of cGAMP MPs and DR2-APM to monocyte-derived DCs, will be tested in co-cultures with autologous T effector cells. Myelin antigen specificity will be determined in Teff and iTreg cells by MHCII tetramer staining.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States